CLINICAL TRIAL: NCT06769971
Title: Phase II Study of Ivonescimab (PD1/VEGF Bispecific) and Cadonilimab（PDL1/CTLA4 Bispecific）in Combination with Etoposide and Carboplatin As First-line Therapy in Patients with Extensive Stage Small Cell Lung Cancer
Brief Title: Phase II Study of Ivonescimab and Cadonilimab in Combination with Chemotherapy in Patients with ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Vice-Director of Cancer Center of West China Hospital, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-AK112-02
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ES-SCLC :Ivonescimab and Cadonilimab plus Chemotherapy (Experimental): Subjects receive Ivonescimab+Cadonilimab + Etoposide+Carboplatin for 4 cycles followed by Ivonescimab and Cadonilimab until progression.
  Interventions: Drug: Ivonescimab; Drug: Cadonilimab; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Ivonescimab — 20mg/kg，IV infusion，Day1，Q3W
Drug: Cadonilimab — 10mg/kg，IV infusion，Day8，Q6W
Drug: Etoposide — 100mg/kg，IV infusion，Day1-3，Q3W
Drug: Carboplatin — AUC 5，IV infusion，Day1，Q3W

SUMMARY:
This is a phase II study. All patients are treatment naive extensive stage small cell lung cancer(ES-SCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of Ivonescimab and Cadonilimab in combination with chemotherapy in patients with ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

1.Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed； 2.18 to 75 years old (at the time of inform consent obtained)； 3.Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1； 4.Have a life expectancy of at least 3 months； 5.Have histologically- or cytologically-confirmed diagnosis of Extensive Stage SCLC； 6.Had not received previous systemic therapy; Or ES-SCLC patients who had received definitive chemoradiotherapy for limited-stage small-cell lung cancer but had disease progression > 6 months earlier; 7.Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator； 8.Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy； 9.Have adequate organ function； 10.All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment；

Exclusion Criteria:

1. Active malignancies within the past 5 years, with the exception of tumors in this study and cured local tumors；
2. Received palliative local treatment, non-specific immunomodulatory treatment within 2 weeks prior to the first dose; and Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 1 weeks prior to the first dose；
3. Subjects who received any prior treatments targeting the mechanism of tumor immunity；
4. Subjects who received any prior anti-angiogenic therapy；
5. Tumor surrounds important blood vessels or has obvious necrosis, cavitation, or invades surrounding important organs and blood vessels；
6. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment；
7. Symptomatic metastases of the central nervous system；
8. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage；
9. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea) within 6 months before the first study drug administration；
10. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
11. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
12. Severe infection within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection that has received systemic anti-infective therapy within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C)；
13. Concurrent enrollment in another clinical study, unless it is a noninterventional clinical study or the follow-up period of the interventional study is more than 4 weeks from the last dose of the prior clinical study or more than 5 half-lives of the prior study drug, whichever is shorter.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 2 years
Safety | Up to approximately 2 years
  Grade 3-4 AEs

SECONDARY OUTCOMES:
DCR | Up to approximately 2 years
DOR | Up to approximately 2 years
TTR | Up to approximately 2 years
PFS | Up to approximately 2 years
OS | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Prof, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China